CLINICAL TRIAL: NCT01788774
Title: Phase I, Open-Label, Randomized, Parallel Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of One Intramuscular Injection of Risperidone ISM® at Different Dose Strengths in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: Pharmacokinetic, Safety, and Tolerability Study of Risperidone ISM® at Different Dose Strengths
Acronym: PRISMA-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROV-RISP-2011-01; 2012-003303-35 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2014-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Pharmacokinetics; Safety; Risperidone ISM®; Intramuscular; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Risperidone ISM 50mg (Other): Three different single doses will be evaluated
  Interventions: Drug: Risperidone ISM 50 mg
- Risperidone ISM 75mg (Other): Three different single doses will be evaluated
  Interventions: Drug: Risperidone ISM 75 mg
- Risperidone ISM 100mg (Other): Three different single doses will be evaluated
  Interventions: Drug: Risperidone ISM 100 mg

INTERVENTIONS:
Drug: Risperidone ISM 50 mg
  Arms: Risperidone ISM 50mg
Drug: Risperidone ISM 75 mg
  Arms: Risperidone ISM 75mg
Drug: Risperidone ISM 100 mg
  Arms: Risperidone ISM 100mg

SUMMARY:
This clinical trial is designed to evaluate different dosages of risperidone ISM, a new long-acting injectable form.

DETAILED DESCRIPTION:
This clinical trial will try to characterize and document the pharmacokinetics of risperidone ISM in schizophrenic or schizoaffective patients after one intramuscular injection at different dose strengths.Likewise, the safety and tolerability of risperidone ISM will be evaluated in the above mentioned population.

Following confirmation of eligibility and a washout period for study-prohibited drugs, a total of 33 subjects will be randomized in a 1:1:1 ratio to receive a single intramuscular (IM) injection of one of the following dosages of study drug:

Group 1: 50 mg risperidone ISM Group 2: 75 mg risperidone ISM Group 3: 100 mg risperidone ISM Several blood samples for plasma pharmacokinetic (PK) assessments will be obtained pre-dose and post-dose. Safety assessments will be conducted at each pre-specified time points.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent.
* Male or female aged ≥ 18 years to < 65 years
* Current diagnosis of schizophrenia or schizoaffective disorder, according to the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders Clinical Trials (SCID-CT) or the DSM-IV-TR
* Medically stable over the last month, and psychiatrically stable without significant symptom exacerbation over the last three months based on the investigator's judgment
* Score of ≤ 4 (moderately ill) on the Clinical Global Impression - Severity of Illness (CGI-S)
* If a sexually active female of childbearing potential, using a medically accepted contraceptive method.

Exclusion Criteria:

* Presence of an uncontrolled, unstable, clinically significant medical condition that in the opinion of the investigator may interfere with the interpretation of safety and PK evaluations
* If female, a positive serum pregnancy test, or planning to become pregnant between now and one month after the last dose of trial medication, or currently breastfeeding a child
* History of neuroleptic malignant syndrome and current or past history of tardive dyskinesia
* Positive urine drug/alcohol screen finding, unless the positive finding can be accounted for by documented prescription use.
* In the investigator's opinion, at imminent risk of committing self-harm
* Use of depot antipsychotics within the last three months
* Receipt of any investigational drugs within the last three months
* Current participation in any other clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve | Pre-dose and 18 time points Post-dose will be carried out within a 75 day time frame

CONTACTS AND LOCATIONS:
Locations (5):
- Zagreb, Croatia
- Russia (2):
  - Moscow
  - Saint Petersburg
- Cape Town, South Africa
- Barcelona, Spain